CLINICAL TRIAL: NCT03204500
Title: A Randomized Clinical Trial, Double Blind, Placebo-controlled of Lithium and Valproate in Amyotrophic Lateral Sclerosis.
Brief Title: Dual Treatment With Lithium and Valproate in ALS.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Principal Investigator, Marie Catherine Boll Woehrlen, MD,PhD, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONACYT234154
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2019-02

CONDITIONS: Amyotrophic Lateral Sclerosis; Amyotrophic Lateral Sclerosis, Sporadic
Keywords: Amyotrophic lateral sclerosis; Dual therapy; Randomized controlled trial; ALSFRS-R
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Amyotrophic lateral sclerosis 1

STUDY DESIGN:
Intervention Model Description: Twenty ALS patients under active treatment vs. twenty ALS patients under placebo treatment. 21 months follow-up whith clinimetry and biomarkers
Who Masked: Participant, Investigator
Masking Description: This is a prospective randomized double-blind placebo-controlled trial. The randomization is made in blocks of 4 treatments (2 active and 2 placebo). Only the 4-digit numbers on the bottle label will identify the type of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment with dual therapy (Experimental): This group is composed by 20 ALS subjects under 600mg valproate and 600 mg of litium carbonate per day, during 21 months. The tablets are given orally with meals.
  Interventions: Combination Product: Active treatment with dual therapy
- placebos (Placebo Comparator): This group is composed by 20 ALS subjects under placebo. Blue tablets ( placebo of VPA) and white tablets (placebo of Li) are administered under the same conditions.
  Interventions: Drug: Placebos

INTERVENTIONS:
Combination Product: Active treatment with dual therapy — Blue pills ( 200 mg of magnesium valproate ) and white pills ( 300 mg of lithium carbonate) are administered orally with meals.
  Arms: Active treatment with dual therapy
Drug: Placebos — Administered orally under the same conditions
  Arms: placebos

SUMMARY:
This is a pilot study in 40 subjects with definite ALS to evaluate the efficacy of valproate and lithium carbonate. After a random assignation of the dual treatment vs. placebo, a follow-up of 20 months will allow to know the clinical and functional evolution so as the status of biomarkers under each treatment.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a rare but fatal condition of the motor neuron. Despite intense therapeutic research in recent years, riluzole remains the only drug with proven efficacy in patients with this disease. In 2008 an Italian clinical-basic study reported benefits with lithium carbonate in both the experimental model of ALS and in a small sample of patients. In the same year, two Chinese studies showed a synergistic neuroprotective effect of valproate administered with lithium in neuronal cultures and in G93A ALS transgenic models.

A clinical trial with lithium carbonate and magnesium valproate,conducted from 2009 to 2012 in 18 patients with diagnostic criteria of ALS compared to a sample of 31 contemporary patients who did not receive the drug showed functionnal stability and an increase in antioxidant defenses in subjects under double treatment. Despite the low level of evidence from this open study, the combination of clinical and biological results as well as the significant increase in survival of treated subjects invites us to conduct a study yielding harsh results on the efficacy of dual treatment.

To obtain harder data, the study will include 40 subjects with random assignation of the treatments (active vs. placebo) by electronic means. The development of the placebo tablets will be in charge of two pharmaceutical companies. Their delivery and purchase will be performed by a nursing team, the same team that will store and conserve the treatments. The preparation and packaging of the tablets for two months for 10 patients will be done regularly in a sterile environment. Two computer engineers will be in charge of the elaboration of the labels and the numerical draw of the treatments. The coordinator of the study will request the treatments in the nursing warehouse equipped with humidity and temperature control. Another person will be trained to make contacts, home deliveries, bottle changes and tablet counts. The appointments will be scheduled by the researchers every 2 months as well as biosecurity exams and magnetic resonance studies in each patient within a 20-month interval.

This pilot study will allow the treatment efficacy to calculate the sample size required for the national and international multicenter clinical trial if relevant, to be promoted at the Mexican Academy of Neurology. It will also allow the study of the behavior of blood and MRI biomarkers ( SOD activity , DTI in cortico-spinal tract, and morphometric indexes).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 40 to 70 years
* of both genders
* female patients who are either postmenopausal for at least 24 months or who are able to practice 2 methods of contraception.
* Clinical diagnosis of definite ALS supported by neurophysiological studies, according to El Escorial reviewed criteria and Awaji criteria.
* Sporadic ALS, a priori.
* Onset of weakness for 1 year ± 6 months
* Vital capacity of at least 60 % of the predicted value
* Other treatment (with riluzole or not) at fixed dosis 2 months before and during all the clinical trial.
* Patients who are willing to give informed consent
* Without gastrostomy
* Without jejunostomy
* Without traqueostomy

Exclusion Criteria:

* Age less than 25 years**
* Patients with uncontrolled diabetes
* Patient with heart failure
* Patient with respiratory vital capacity < 60%
* Hepatic failure
* Dysthyroidism
* Do not give or sign informed consent
* Women in lactation, pregnancy or possibility of pregnancy
* Patients with significant sensory abnormalities and uncompensated medical illnesses
* Laboratory abnormalities consistent with clinically significant cardiovascular, respiratory, haematological, metabolic, hepatic and renal disease.
* Patients with gastrostomy
* With jejunostomy
* With nasogastric tube
* Tracheotomy and invasive ventilation
* Treatment with investigational drug within 3 months prior to screening

  * Patients aged 26 to 39 years can be included at the discretion of medical researchers.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Changes in ALSFRS-R | Every 2 months for 20 months
  To evaluate the effect of VPA+Li on progression of ALS by measuring functionnal changes from baseline in ALSFRS-R.

SECONDARY OUTCOMES:
Changes in score in ALSAQ-5 | Baseline, Month 10, Month 20
  Changes from baseline in ALSAQ-5, a brief self-administered quality of life scale.
Changes from baseline in FA (fractional anisotropy) | Baseline and month18
  DTI biomarkers in corticospinal tract are measured in 6 regions bilaterally

CONTACTS AND LOCATIONS:
Overall Officials: MARIE CATHERINE BOLL, MD,PhD., Principal Investigator — 525556063822
Locations (1):
- Instituto Nacional de Neurologia Y Neurocirugia Mvs, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boll MC, Bayliss L, Vargas-Canas S, Burgos J, Montes S, Penaloza-Solano G, Rios C, Alcaraz-Zubeldia M. Clinical and biological changes under treatment with lithium carbonate and valproic acid in sporadic amyotrophic lateral sclerosis. J Neurol Sci. 2014 May 15;340(1-2):103-8. doi: 10.1016/j.jns.2014.03.005. Epub 2014 Mar 11. PMID 24667005
- [Background] Boll MC, Alcaraz-Zubeldia M, Montes S, Murillo-Bonilla L, Rios C. Raised nitrate concentration and low SOD activity in the CSF of sporadic ALS patients. Neurochem Res. 2003 May;28(5):699-703. doi: 10.1023/a:1022853531855. PMID 12716019
- [Background] Caldero J, Brunet N, Tarabal O, Piedrafita L, Hereu M, Ayala V, Esquerda JE. Lithium prevents excitotoxic cell death of motoneurons in organotypic slice cultures of spinal cord. Neuroscience. 2010 Feb 17;165(4):1353-69. doi: 10.1016/j.neuroscience.2009.11.034. Epub 2009 Nov 22. PMID 19932742
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Chen RW, Chuang DM. Long term lithium treatment suppresses p53 and Bax expression but increases Bcl-2 expression. A prominent role in neuroprotection against excitotoxicity. J Biol Chem. 1999 Mar 5;274(10):6039-42. doi: 10.1074/jbc.274.10.6039. PMID 10037682
- [Background] Feng HL, Leng Y, Ma CH, Zhang J, Ren M, Chuang DM. Combined lithium and valproate treatment delays disease onset, reduces neurological deficits and prolongs survival in an amyotrophic lateral sclerosis mouse model. Neuroscience. 2008 Aug 26;155(3):567-72. doi: 10.1016/j.neuroscience.2008.06.040. Epub 2008 Jun 21. PMID 18640245
- [Background] Fornai F, Longone P, Cafaro L, Kastsiuchenka O, Ferrucci M, Manca ML, Lazzeri G, Spalloni A, Bellio N, Lenzi P, Modugno N, Siciliano G, Isidoro C, Murri L, Ruggieri S, Paparelli A. Lithium delays progression of amyotrophic lateral sclerosis. Proc Natl Acad Sci U S A. 2008 Feb 12;105(6):2052-7. doi: 10.1073/pnas.0708022105. Epub 2008 Feb 4. PMID 18250315
- [Background] Kimura F, Fujimura C, Ishida S, Nakajima H, Furutama D, Uehara H, Shinoda K, Sugino M, Hanafusa T. Progression rate of ALSFRS-R at time of diagnosis predicts survival time in ALS. Neurology. 2006 Jan 24;66(2):265-7. doi: 10.1212/01.wnl.0000194316.91908.8a. PMID 16434671
- [Background] Leng Y, Liang MH, Ren M, Marinova Z, Leeds P, Chuang DM. Synergistic neuroprotective effects of lithium and valproic acid or other histone deacetylase inhibitors in neurons: roles of glycogen synthase kinase-3 inhibition. J Neurosci. 2008 Mar 5;28(10):2576-88. doi: 10.1523/JNEUROSCI.5467-07.2008. PMID 18322101
- [Background] Machado Ximenes JC, Lima Verde EC, Naffah-Mazzacoratti MG, Barros Viana GS. Valproic Acid, a Drug with Multiple Molecular Targets Related to Its Potential Neuroprotective Action. Neuroscience & Medicine, 2012, 3, 107-123 http://dx.doi.org/10.4236/nm.2012.31016
- [Background] Yasuda S, Liang MH, Marinova Z, Yahyavi A, Chuang DM. The mood stabilizers lithium and valproate selectively activate the promoter IV of brain-derived neurotrophic factor in neurons. Mol Psychiatry. 2009 Jan;14(1):51-9. doi: 10.1038/sj.mp.4002099. Epub 2007 Oct 9. PMID 17925795
- [Background] Jenkinson C, Fitzpatrick R. Reduced item set for the amyotrophic lateral sclerosis assessment questionnaire: development and validation of the ALSAQ-5. J Neurol Neurosurg Psychiatry. 2001 Jan;70(1):70-3. doi: 10.1136/jnnp.70.1.70. PMID 11118250